CLINICAL TRIAL: NCT03173417
Title: Safety and Efficacy Evaluation of IM19 CAR-T Cells On CD19+ Refractory or Relapsed B-ALL Patients
Brief Title: Safety and Efficacy Evaluation of IM19 CAR-T Cells (IM19CAR-T)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMCART201702
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM19 CART (Experimental): All patients will be treated with fludarabine and cyclophosphamide for 3 days,then,CAR-T cells expressing CD19 CAR will be infused 24-96 hours later.
  Interventions: Biological: IM19 CAR-T; Drug: fludarabine and cyclophosphamide

INTERVENTIONS:
Biological: IM19 CAR-T — T Cells Expressing an Anti-CD19 Chimeric Antigen Receptor
  Other Names: IM19
Drug: fludarabine and cyclophosphamide — Two days before cell infusion,all patients will be treated with fludarabine and cyclophosphamide for 3 days
  Other Names: FC

SUMMARY:
Assessment of the Safety and Feasibility of Administering T Cells Expressing an Anti-CD19 Chimeric Antigen Receptor to Patients With CD19+ B-cell leukemia.

DETAILED DESCRIPTION:
Assessment of the Safety and Feasibility of Administering T Cells Expressing an Anti-CD19 Chimeric Antigen Receptor to Patients With CD19+ B-cell leukemia and determine the best dosage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CD19+ Refractory or Relapsed B-ALL（At least 2 prior combination chemotherapy regimens）
2. To be aged 3 to 75 years
3. Blast in blood ≤ 30%
4. ECOG score ≤2
5. Women of childbearing potential must have a urine pregnancy test taken and proven negative prior to the treatment. All patients agree to use reliable methods of contraception during the trial period and until follow-up for the last time.
6. Voluntary participation in the clinical trials and sign the informed consent.

Exclusion Criteria:

1. Intracranial hypertension or unconsciousness
2. Respiratory failure
3. CD19 negative
4. Disseminated intravascular coagulation
5. ALT /AST>3 x normal value; Creatinine> 1.5 x normal value; Bilirubin >2.0 x normal value
6. Hematosepsis or Uncontrolled active infection
7. Uncontrolled diabetes
8. Abalienation;
9. WHO Sscore >3
10. Patients in pregnancy or breast-feeding period
11. Previously treatment with any gene therapy products
12. Any uncontrolled medical disorders that the researchers consider are not eligible to participate the clinical trial
13. Any situation that would increase dangerousness of subjects or disturb the outcome of the clinical study according to the researcher's evaluation.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | 2 years
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment Adverse events assessed according to NCI-CTCAE v4.0 criteria 2.

SECONDARY OUTCOMES:
Overall response rate | 2 years
  An objective response is defined as: (1) a morphologic complete response (CR) or (2) a complete response with incomplete recovery of counts (CRi) (based on NCCN guidelines (National Comprehensive Cancer Network (NCCN), 2014) or (3) a negative minimal residual disease assessed by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: PEIHUA LU, MD, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen M, Fu M, Wang A, Wu X, Zhen J, Gong M, Zhang X, Yue G, Du Q, Zhao W, Zhao Y, Lu P, Wang H. Cytoplasmic CD79a is a promising biomarker for B lymphoblastic leukemia follow up post CD19 CAR-T therapy. Leuk Lymphoma. 2022 Feb;63(2):426-434. doi: 10.1080/10428194.2021.1980214. Epub 2021 Oct 21. PMID 34672246
- [Derived] Zhang X, Lu XA, Yang J, Zhang G, Li J, Song L, Su Y, Shi Y, Zhang M, He J, Song D, Lv F, Li W, Wu Y, Wang H, Liu H, Zhou X, He T, Lu P. Efficacy and safety of anti-CD19 CAR T-cell therapy in 110 patients with B-cell acute lymphoblastic leukemia with high-risk features. Blood Adv. 2020 May 26;4(10):2325-2338. doi: 10.1182/bloodadvances.2020001466. PMID 32453841